CLINICAL TRIAL: NCT07155317
Title: The TIME Trial - Phase II Randomized Controlled Trial of Time-of-Day Specified Immunotherapy for Advanced Melanoma
Brief Title: Time-of-Day Specified Immunotherapy for Advanced Melanoma, The TIME Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Lowe, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008806; NCI-2025-03025 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00008806 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP6451-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2025-08-21; First posted 2025-09-04 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced Acral Melanoma; Advanced Cutaneous Melanoma; Advanced Mucosal Melanoma; Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Acral Melanoma; Metastatic Cutaneous Melanoma; Metastatic Mucosal Melanoma; Unresectable Acral Melanoma; Unresectable Cutaneous Melanoma; Unresectable Mucosal Melanoma
MeSH Terms: conditions — Melanoma | interventions — Biopsy; Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes at 0800-1100 on day 1 of each cycle. Cycles repeat every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance nivolumab for up to a total of 2 years. Patients wear an actigraphy device for 5-7 days at enrollment prior to first infusion and for up to 4 weeks then over 3 weeks starting with visit 4. Patients also undergo check swab and blood sample collection, CT or MRI and MRI or CT of brain throughout the study. Additionally, patients may optionally undergo tumor tissue biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Other: Medical Device Usage and Evaluation; Biological: Nivolumab; Other: Questionnaire Administration
- Arm II (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes at 1100-1400 on day 1 of each cycle. Cycles repeat every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance nivolumab for up to a total of 2 years. Patients wear an actigraphy device for 5-7 days at enrollment prior to first infusion and for up to 4 weeks then over 3 weeks starting with visit 4. Patients also undergo check swab and blood sample collection, CT or MRI and MRI or CT of brain throughout the study. Additionally, patients may optionally undergo tumor tissue biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Other: Medical Device Usage and Evaluation; Biological: Nivolumab; Other: Questionnaire Administration
- Arm III (nivolumab, ipilimumab) (Active Comparator): Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes at 1400-1700 on day 1 of each cycle. Cycles repeat every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance nivolumab for up to a total of 2 years. Patients wear an actigraphy device for 5-7 days at enrollment prior to first infusion and for up to 4 weeks then over 3 weeks starting with visit 4. Patients also undergo check swab and blood sample collection, CT or MRI and MRI or CT of brain throughout the study. Additionally, patients may optionally undergo tumor tissue biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Other: Medical Device Usage and Evaluation; Biological: Nivolumab; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo check swab and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Medical Device Usage and Evaluation — Wear an actigraphy device
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests the safety and effectiveness of giving ipilimumab and nivolumab in the morning compared to other times of day in treating patients with melanoma that is stage IV or that cannot be removed by surgery (unresectable). Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the tumor and may interfere with the ability of tumor cells to grow and spread. While some patients have impressive outcomes with both of these drugs, over 40% of patients do not experience any clinical benefit. Studies have shown that the time of day that vaccines and other therapies are given have had an impact on response and survival. It is not known, however, whether time of day has an impact on response to immune checkpoint inhibitors, such as ipilimumab and nivolumab. Giving ipilimumab and nivolumab earlier in the day compared to later in the day may improve response to treatment and survival in patients with stage IV or unresectable melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the progression-free survival (PFS) following administration of immunotherapy at different time-of-day intervals for previously untreated unresectable or metastatic melanoma.

SECONDARY OBJECTIVES:

I. To compare adverse events (AEs). II. Rate of receiving all immunotherapy doses as scheduled. III. Objective response rate. IV. Melanoma specific survival (MSS) and overall survival (OS). V. Patient-reported quality of life (QOL).

TERTIARY/EXPLORATORY OBJECTIVE:

I. To explore immune biomarkers associated with clinical efficacy (PFS, OS).

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive nivolumab intravenously (IV) over 60 minutes and ipilimumab IV over 90 minutes at 0800-1100 on day 1 of each cycle. Cycles repeat every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance nivolumab for up to a total of 2 years. Patients wear an actigraphy device for 5-7 days at enrollment prior to first infusion and for up to 4 weeks then over 3 weeks starting with visit 4. Patients also undergo check swab and blood sample collection, computed tomography (CT) or magnetic resonance imaging (MRI) and MRI or CT of brain throughout the study. Additionally, patients may optionally undergo tumor tissue biopsy throughout the study.

ARM II: Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes at 1100-1400 on day 1 of each cycle. Cycles repeat every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance nivolumab for up to a total of 2 years. Patients wear an actigraphy device for 5-7 days at enrollment prior to first infusion and for up to 4 weeks then over 3 weeks starting with visit 4. Patients also undergo check swab and blood sample collection, CT or MRI and MRI or CT of brain throughout the study. Additionally, patients may optionally undergo tumor tissue biopsy throughout the study.

ARM III: Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes at 1400-1700 on day 1 of each cycle. Cycles repeat every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance nivolumab for up to a total of 2 years. Patients wear an actigraphy device for 5-7 days at enrollment prior to first infusion and for up to 4 weeks then over 3 weeks starting with visit 4. Patients also undergo check swab and blood sample collection, CT or MRI and MRI or CT of brain throughout the study. Additionally, patients may optionally undergo tumor tissue biopsy throughout the study.

After completion of study treatment, patients are followed up every 3 months for 12 months, then for up to year 5.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed American Joint Committee on Cancer (AJCC) 8th edition stage IV unresectable cutaneous, acral, or mucosal melanoma
* No uveal melanoma
* Patients with asymptomatic, non-hemorrhagic brain metastases < 2 cm are eligible
* No prior immunotherapy within 1 year, (serine/threonine-protein kinase B-raf [BRAF]/mitogen-activated protein kinase [MEK] inhibitors allowed)
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Age ≥ 18
* Adequate organ function to receive ipilimumab/nivolumab

Exclusion Criteria:

* Immunosuppression (> 10mg prednisone daily)
* Active autoimmune disease that would preclude the administration of immunotherapy
* Active leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) A versus (vs.) C and B vs. C | From randomization to progression or death, assessed up to 5 years
  Will be determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Will be compared between arms with a log rank test. The hazard ratio and the corresponding 95% confidence interval (CI) for the A vs. C and B vs. C comparisons will be estimated in a Cox proportional hazards model using the randomized arm as a single covariate. The PFS curves for each randomized arm will be estimated using the Kaplan-Meier (KM) method. In addition, PFS rates at specific time points will be estimated using KM estimates on the PFS curve for each randomized arm. Associated 2-sided 95% CIs will be calculated using the Greenwood formula (using log-log transformation).

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events (AE) | Up to 100 days after last dose of study treatment
  Will be determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5. Frequencies and percentages will be used to summarize safety events. All treatment-associated AE event rates, as well as treatment-associated grade 3 or higher AE event rates will be reported. Event rates will be compared between arms using a Chi-square test. Differences in event rates will be reported, and 95% CIs will be estimated.
Objective Response Rate (ORR) | Up to 3 months
  Will be defined as complete response and/or partial response assessed using RECIST 1.1 criteria. Will be estimated as a proportion, with an exact 95% CI estimated using the Clopper-Pearson method. ORR will be compared between arms using a Chi-square test.
Overall Survival (OS) | From randomization to death from any cause, assessed up to 5 years
  Will be compared between arms with a log rank test. The hazard ratio and the corresponding 95% CIs for the A vs. C and B vs. C comparisons will be estimated in a Cox proportional hazards model using the randomized arm as a single covariate. The OS curves for each randomized arm will be estimated using the KM method. In addition, OS rates at specific time points will be estimated using KM estimates on the OS curve for each randomized arm. Associated 2-sided 95% CIs will be calculated using the Greenwood formula (using log-log transformation).
PFS A vs. B | From randomization to progression or death, assessed up to 5 years
  Will be determined using RECIST 1.1. PFS will be compared between arms with a log rank test. The hazard ratio and the corresponding 95% CI for the A vs. B comparison will be estimated in a Cox proportional hazards model using the randomized arm as a single covariate. The PFS curves for each randomized arm will be estimated using the KM method. In addition, PFS rates at specific time points will be estimated using KM estimates on the PFS curve for each randomized arm. Associated 2-sided 95% CIs will be calculated using the Greenwood formula (using log-log transformation).
Disease Specific Survival | Up to 5 years
  To explore immune biomarkers associated with clinical efficacy from the pre-treatment and post-treatment melanoma biopsy specimens and peripheral blood.
Rate of Receiving all Immunotherapy Doses as Scheduled | Up to 4 cycles (cycle length = 3 weeks)
  To compare rate of receiving all immunotherapy doses as scheduled, of subjects with previously untreated unresectable or metasatic melanoma who receive immunotherapy infusions at different time-of-day intervals, and impact of quality of life on timing of infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lowe, MD, MA, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia